CLINICAL TRIAL: NCT00365976
Title: Double-blind, Placebo-controlled Study of the Safety and Efficacy of Eszopiclone in the Treatment of Insomnia in Patients With Chronic Low Back Pain
Brief Title: Study of the Insomnia in Patients With Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00011697; ESRC 032
Record Dates: First submitted 2006-08-16; First posted 2006-08-18 (Estimated); Results first posted 2013-06-07 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-06

CONDITIONS: Primary Insomnia
Keywords: Insomnia; Low Back Pain; Hypnotics; Eszopiclone; Pain; Disability
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Low Back Pain; Pain | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Active Comparator): Eszopiclone
  Interventions: Drug: Eszopiclone

INTERVENTIONS:
Drug: Eszopiclone — Eszopiclone 3 mg po nightly for duration of study blind phase.
  Other Names: Lunesta
  Arms: 2
Drug: Placebo — Placebo nightly over duration of double blind study phase
  Arms: 1

SUMMARY:
The purpose of this study is to examine whether insomnia due to chronic low back pain can improve with use of eszopiclone.

DETAILED DESCRIPTION:
There is a great need to develop effective treatments for insomnia in patients with chronic low-back pain. Chronic low-back pain is among the most prevalent of all health complaints, is associated with enormous health-care and productivity costs, reduced quality of life, and limitation of function and is almost universally associated with insomnia (Rives and Douglas, 2004). While it had long been believed that insomnia was a symptom of pain conditions and of little consequence in its' own right, a growing literature suggests that insomnia has important effects on the clinical course of pain syndromes (Smith and Haythornthwaite, 2004). While pain may disrupt sleep, it appears that problems with sleep increase pain and are associated with impairments in daytime function. The emerging point of view is that specific treatment for both pain and insomnia is needed for optimal clinical management (Smith and Haythornthwaite, 2004). Surprisingly, despite the fact that chronic low-back pain is the most common pain condition, the treatment of insomnia in this disease has never been studied. As a result, we propose to carry out the first double-blind placebo-controlled study of the treatment insomnia in patients with chronic low back pain.

Comparison(s): We will test the hypothesis that treating the insomnia with eszopiclone 3 mg (ESZ) along with management of pain with naproxen 500 mg bid (NAP) will result in statistically significantly improved sleep compared with placebo. We also propose to test as a secondary hypothesis that treatment with ESZ will lead to significant improvement in pain and daytime function vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of insomnia based on DSM-IV criteria for insomnia due to a general medical condition (low-back pain);

  * The insomnia must not predate the onset of low-back pain by more than 1 month;
  * Usual nightly TST (Total Sleep Time) < 6.5 hours and/or usual SOL (Sleep Onset Latency) > 30 minutes for the last month prior to screening;
  * ISI (Insomnia Severity Index) > 14 (at least moderate insomnia);
  * Age 21-64 years;
  * Greater than 40 on VAS (Visual Analog Scale) for pain (scale is 0-no pain to 100-worst imaginable pain);
  * Patient Global Impression of Pain of at least 3 (on a 1-5 scale, indicating at least moderate severity);
  * reported Back pain must be greater than reported leg pain, and there must be no signs of spinal nerve root compression;
  * presence of normal motor strength on exam;
  * duration of chronic low back pain of greater than three months;
  * low back pain location must be inferior to T12 and superior to the gluteal fold.

Exclusion Criteria:

* • Significant medical or neurological illness in excess of that which is directly responsible for the chronic low back pain;

  * the presence of an active and significant psychiatric disease with a substantive impact on sleep;
  * meeting DSM-IV criteria for an Axis I disorder within the last three months, or meeting criteria for substance abuse within the last 12 months;
  * current pregnancy; history of hypersensitivity, intolerance, or contraindication to Naproxen/Lansoprazole or Eszopiclone;
  * baseline creatinine of 2.0 or greater; patient taking other medications having significant renal effects (e.g. lithium, ACE inhibitor, angiotensin receptor antagonist, or thiazide/loop diuretics);
  * patients taking other anticoagulants; patients having an allergy to aspirin; history of diagnosed gastric or duodenal ulcer;
  * history of bleeding or clotting diathesis; lifetime history of myocardial infarction or cerebrovascular accident;
  * Elevated PT/PTT/INR (Prothrombin Time, Partial Thromboplastin Time, International Normalized Ratio)at screening;
  * Abnormal kidney function detected in screening labs;
  * history of back related surgery within the past 3 months; history of corticosteroid use in the past 30 days;
  * presence of currently pending litigation or worker's compensation claim related to the chronic low back pain;
  * inability to follow study procedures or complete the study; or the use of any medications that could affect sleep within 5 half-lives of screening;
  * history of back surgery within the past 2 years with the exception of a discectomy;
  * pregnant or lactating females;
  * women of child-bearing potential who will not agree to use approved means of birth control during the trial;
  * history of any surgery within the past one month; history of any major physical trauma within the last 6 months;
  * history of corticosteroid use within the last 90 days; diagnosis of rheumatoid or psoriatic arthritis;
  * history of fibromyalgia;
  * presence of spondyloarthropathy;
  * presence of sciatica;
  * spinal stenosis;
  * presence of any vertebral fractures, spondylolisthesis; or radicular back pain.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2006-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Krystal, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Berry H, Bloom B, Hamilton EB, Swinson DR. Naproxen sodium, diflunisal, and placebo in the treatment of chronic back pain. Ann Rheum Dis. 1982 Apr;41(2):129-32. doi: 10.1136/ard.41.2.129. PMID 6462116
- [Background] Benca RM, Ancoli-Israel S, Moldofsky H. Special considerations in insomnia diagnosis and management: depressed, elderly, and chronic pain populations. J Clin Psychiatry. 2004;65 Suppl 8:26-35. PMID 15153065
- [Background] Coats TL, Borenstein DG, Nangia NK, Brown MT. Effects of valdecoxib in the treatment of chronic low back pain: results of a randomized, placebo-controlled trial. Clin Ther. 2004 Aug;26(8):1249-60. doi: 10.1016/s0149-2918(04)80081-x. PMID 15476906
- [Background] Curran MP, Wellington K. Delayed-release lansoprazole plus naproxen. Drugs. 2004;64(17):1915-9; discussion 1920-1. doi: 10.2165/00003495-200464170-00008. PMID 15329041
- [Background] Edinger JD, Means MK, Stechuchak KM, Olsen MK. A pilot study of inexpensive sleep-assessment devices. Behav Sleep Med. 2004;2(1):41-9. doi: 10.1207/s15402010bsm0201_4. PMID 15600223
- [Background] Hagg O, Fritzell P, Nordwall A; Swedish Lumbar Spine Study Group. The clinical importance of changes in outcome scores after treatment for chronic low back pain. Eur Spine J. 2003 Feb;12(1):12-20. doi: 10.1007/s00586-002-0464-0. Epub 2002 Oct 24. PMID 12592542
- [Background] Holm I, Friis A, Storheim K, Brox JI. Measuring self-reported functional status and pain in patients with chronic low back pain by postal questionnaires: a reliability study. Spine (Phila Pa 1976). 2003 Apr 15;28(8):828-33. PMID 12698128
- [Background] Katz N, Rodgers DB, Krupa D, Reicin A. Onset of pain relief with rofecoxib in chronic low back pain: results of two four-week, randomized, placebo-controlled trials. Curr Med Res Opin. 2004 May;20(5):651-8. doi: 10.1185/030079904125003160. PMID 15140330
- [Background] Koes BW, Scholten RJ, Mens JM, Bouter LM. Efficacy of non-steroidal anti-inflammatory drugs for low back pain: a systematic review of randomised clinical trials. Ann Rheum Dis. 1997 Apr;56(4):214-23. doi: 10.1136/ard.56.4.214. PMID 9165992
- [Background] Krystal AD, Walsh JK, Laska E, Caron J, Amato DA, Wessel TC, Roth T. Sustained efficacy of eszopiclone over 6 months of nightly treatment: results of a randomized, double-blind, placebo-controlled study in adults with chronic insomnia. Sleep. 2003 Nov 1;26(7):793-9. doi: 10.1093/sleep/26.7.793. PMID 14655910
- [Background] Lai KC, Lam SK, Chu KM, Hui WM, Kwok KF, Wong BC, Hu HC, Wong WM, Chan OO, Chan CK. Lansoprazole reduces ulcer relapse after eradication of Helicobacter pylori in nonsteroidal anti-inflammatory drug users--a randomized trial. Aliment Pharmacol Ther. 2003 Oct 15;18(8):829-36. doi: 10.1046/j.1365-2036.2003.01762.x. PMID 14535877
- [Background] Luo X, Pietrobon R, Curtis LH, Hey LA. Prescription of nonsteroidal anti-inflammatory drugs and muscle relaxants for back pain in the United States. Spine (Phila Pa 1976). 2004 Dec 1;29(23):E531-7. doi: 10.1097/01.brs.0000146453.76528.7c. PMID 15564901
- [Background] Ostelo RW, de Vet HC. Clinically important outcomes in low back pain. Best Pract Res Clin Rheumatol. 2005 Aug;19(4):593-607. doi: 10.1016/j.berh.2005.03.003. PMID 15949778
- [Background] Pallay RM, Seger W, Adler JL, Ettlinger RE, Quaidoo EA, Lipetz R, O'Brien K, Mucciola L, Skalky CS, Petruschke RA, Bohidar NR, Geba GP. Etoricoxib reduced pain and disability and improved quality of life in patients with chronic low back pain: a 3 month, randomized, controlled trial. Scand J Rheumatol. 2004;33(4):257-66. doi: 10.1080/03009740410005728. PMID 15370723
- [Background] Rives PA, Douglass AB. Evaluation and treatment of low back pain in family practice. J Am Board Fam Pract. 2004 Nov-Dec;17 Suppl:S23-31. doi: 10.3122/jabfm.17.suppl_1.s23. PMID 15575027
- [Background] Smith MT, Haythornthwaite JA. How do sleep disturbance and chronic pain inter-relate? Insights from the longitudinal and cognitive-behavioral clinical trials literature. Sleep Med Rev. 2004 Apr;8(2):119-32. doi: 10.1016/S1087-0792(03)00044-3. PMID 15033151
- [Background] Zammit GK, McNabb LJ, Caron J, Amato DA, Roth T. Efficacy and safety of eszopiclone across 6-weeks of treatment for primary insomnia. Curr Med Res Opin. 2004 Dec;20(12):1979-91. doi: 10.1185/174234304x15174. PMID 15701215
- [Derived] Goforth HW, Preud'homme XA, Krystal AD. A randomized, double-blind, placebo-controlled trial of eszopiclone for the treatment of insomnia in patients with chronic low back pain. Sleep. 2014 Jun 1;37(6):1053-60. doi: 10.5665/sleep.3760. PMID 24882900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy adult volunteers with low back pain who met diagnostic criteria for insomnia were recruited through newspaper advertisements, posted announcements and physician referrals. Of those 70, 10 did not meet inclusion criteria, and 2 chose not to participate. The remaining 58 were randomized.
Pre-assignment Details: Qualifying subjects were switched from their current pain regimen to naproxen and lansoprazole. We excluded those with: significant medical or neurological illness other than LBP; psychiatric disease impacting sleep; substance abuse; history of hypersensitivity or contraindication to NAP/LAN or ESZ; abnormalities on baseline laboratory tests.
Groups:
- Eszopiclone: Eszopiclone : Eszopiclone 3 mg po nightly for duration of study blind phase.
- Placebo: Placebo : Placebo nightly over duration of double blind study phase.
Period: Overall Study
Arm/Group | Eszopiclone | Placebo
Started | 33 | 25
Completed | 32 | 20
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eszopiclone | Placebo | Total
Number analyzed (Participants) | 33 | 25 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 25 | 58
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (11.0) | 40.1 (12.8) | 43.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 13 | 7 | 20
Region of Enrollment [Number; unit: participants]
  United States | 33 | 25 | 58

OUTCOME MEASURES:

1. Primary Outcome: Mean Subjective Sleep Diary Derived Total Sleep Time (TST)
Description: Nightly total sleep time was averaged from diary entries.
Time Frame: Postnaprosyn baseline, Week 1, week 2, week 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 32 | 20
Minutes
  postnaprosyn baseline | 316.96 (91.55) | 380.45 (81.33)
  week 1 | 403.47 (77.67) | 375.56 (88.74)
  week 2 | 421.97 (68.28) | 382.11 (96.13)
  Week 4 | 411.97 (66.87) | 388.96 (99.02)

2. Secondary Outcome: Visual Analog Scale Pain Ratings (VAS)
Description: Scores are measured on a 100 mm Visual Analog Scale (VAS). The VAS scale ranges from 0 to 100 mm with the lower score indicating less pain and the higher score indicating greater pain
Time Frame: Postnaprosyn baseline, Week 1, Week 2, Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 32 | 20
units on a scale
  Postnaprosyn Baseline | 48.51 (16.22) | 53.79 (20.96)
  Week 1 | 40.72 (17.13) | 51.99 (20.83)
  Week 2 | 34.70 (18.49) | 51.25 (19.61)
  Week 4 | 31.69 (17.92) | 51.60 (22.44)

3. Secondary Outcome: Mean Sleep Onset Latency (SOL)
Time Frame: Postnaprosyn Baseline, Week 1, Week 2 week 4
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 32 | 20
minutes
  Postnaprosyn Baseline | 38.28 (23.90) | 34.11 (25.93)
  Week 1 | 22.36 (16.59) | 27.00 (18.28)
  Week 2 | 17.50 (12.33) | 23.10 (19.68)
  Week 4 | 15.28 (12.95) | 19.91 (12.30)

4. Secondary Outcome: Wake Time After Sleep Onset
Time Frame: Postnaprosyn Baseline, Week 1, Week 2 week 4
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 32 | 20
minutes
  Postnaprosyn Baseline | 91.51 (55.91) | 81.43 (54.58)
  Week 1 | 49.34 (32.62) | 76.71 (65.84)
  Week 2 | 37.07 (22.21) | 81.32 (76.30)
  Week 4 | 36.74 (28.44) | 76.18 (65.50)

5. Secondary Outcome: Number of Awakenings
Time Frame: Postnaprosyn Baseline, Week 1, Week 2 week 4
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 32 | 20
awakenings
  Postnaprosyn Baseline | 2.29 (1.48) | 2.08 (1.51)
  Week 1 | 1.31 (1.02) | 1.98 (1.43)
  Week 2 | 1.35 (0.99) | 2.13 (1.81)
  Week 4 | 1.33 (1.01) | 2.34 (1.79)

6. Secondary Outcome: Sleep Quality Ratings
Description: Sleep quality ratings are based on a 1-10 Likert scale. Low scores represent poorer sleep quality and higher scores represent better quality sleep
Time Frame: Postnaprosyn Baseline, Week 1, Week 2 week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 32 | 20
units on a scale
  Postnaprosyn Baseline | 4.52 (1.45) | 4.44 (1.66)
  Week 1 | 5.99 (1.43) | 4.90 (1.83)
  Week 2 | 6.18 (1.45) | 5.33 (1.77)
  Week 4 | 6.38 (1.66) | 5.29 (2.00)

7. Secondary Outcome: Insomnia Severity Index (ISI)
Description: The ISI is a seven-item self-report questionnaire that provides a global measure of insomnia severity based on difficulty falling or staying asleep, satisfaction with sleep, or degree of impairment with daytime functioning. The total score ranges from 0-28: 0-7 (no clinical insomnia), 8-14 (subthreshold insomnia), 15-21 (insomnia of moderate severity), and 22-28 (severe insomnia).
Time Frame: Prenaprosyn Baseline, Postnaprosyn Baseline, Week 1, Week 2 week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 32 | 20
units on a scale
  Prenaprosyn Baseline | 18.85 (4.01) | 20.26 (4.07)
  Postnaprosyn baseline | 18.00 (3.41) | 16.78 (4.32)
  Week 1 | 11.28 (6.10) | 12.85 (5.97)
  Week 2 | 10.61 (6.60) | 12.74 (6.39)
  Week 4 | 8.38 (6.42) | 13.75 (6.78)

8. Secondary Outcome: Patient Global Impression of Pain Ratings
Description: Pain ratings included a global impression of pain rating (PGI) (1-5 rating with 1 being little pain and 5 is worst pain)
Time Frame: postnaprosyn Baseline, Week 1, Week 2 week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 32 | 20
units on a scale
  postnaprosyn Baseline | 4.02 (0.95) | 3.90 (1.47)
  Week 1 | 3.54 (1.17) | 3.82 (1.45)
  Week 2 | 3.30 (1.27) | 4.01 (1.12)
  Week 4 | 3.08 (1.28) | 3.80 (1.14)

9. Secondary Outcome: Roland Morris Low Back Pain Inventory (RMLBPI)
Description: The Roland-Morris Low Back Pain Disability Questionnaire (RMLBPDQ) is a 24-item instrument that assesses the extent to which activities of daily living are affected by LBP. It is composed of 24 "yes-no" items assessing potential disabilities.
  Scores range from 0 (no disability) to 24 (severe disability).
Time Frame: prenaprosyn baseline, postnaprosyn Baseline, Week 1, Week 2, week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 32 | 20
units on a scale
  prenaprosyn Baseline | 12.27 (5.70) | 11.33 (5.66)
  postnaprosyn Baseline | 9.97 (5.55) | 10.30 (5.75)
  Week 1 | 9.10 (6.37) | 9.05 (6.32)
  Week 2 | 7.63 (6.34) | 9.32 (6.25)
  Week 4 | 6.59 (5.49) | 7.94 (6.99)

10. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D-24)
Description: The Hamilton Depression Scale - 24 Items (HAM-D-24) measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 76. The higher the score, the more severe.
Time Frame: prenaprosyn baseline, postnaprosyn Baseline, Week 1, Week 2, week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 32 | 20
units on a scale
  prenaprosyn Baseline | 6.45 (2.26) | 7.10 (3.83)
  postnaprosyn Baseline | 6.38 (2.37) | 6.57 (3.63)
  Week 1 | 4.54 (3.71) | 5.53 (3.28)
  Week 2 | 4.14 (3.50) | 5.07 (3.61)
  Week 4 | 2.62 (2.61) | 6.21 (5.18)

11. Secondary Outcome: Short Form 36 Health Survey Questionnaire (SF-36)
Description: The SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The vitality sub-score assesses energy and fatigue, and ranges from 0 (worst) - 100 (best).
Time Frame: Baseline, week 1, week 2, week 4
Population: Data not collected.
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: State-Trait Anxiety Inventory (STAI)
Description: Self-rating assessment of anxiety measured by STAI, state anxiety inventory (Scale 40-160, where a lower value shows a larger improvement)
Time Frame: Baseline, week 1, week 2, week 4
Population: Data not collected.
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Eszopiclone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/25
Other Adverse Events (participants affected / at risk) | 0/33 | 0/25

LIMITATIONS AND CAVEATS:
1. We obtained only self-reported sleep outcomes.
2. The period of double-blind treatment was relatively short.
3. We excluded all subjects who might have required opioid therapy to manage their pain which limits study generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less